CLINICAL TRIAL: NCT05440006
Title: Randomized, Open, Two Cycle, Two Sequence, Cross Reference Designed Study on the Effect of Food on the Pharmacokinetics of Fuzuloparib Capsules in Chinese Healthy Adult Subjects
Brief Title: A Study of Food Effect on the Pharmacokinetics of Fuzuloparib Capsules in Chinese Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR3162-I-122
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: There will be 20 volunteers to receive the treatment, and each treatment will be followed by 72 hours of blood sampling for pharmacokinetic and safety.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fed+ Fasted (Experimental): The first cycle with high-fat meal, the second cycle under fasting.
  Interventions: Drug: Fuzuloparib
- Fasted + Fed (Experimental): The first cycle under fasting, the second cycle with high-fat meal.
  Interventions: Drug: Fuzuloparib

INTERVENTIONS:
Drug: Fuzuloparib — Fuzuloparib Capsules; 150mg; single dose per cycle.

SUMMARY:
The objective of the study is to assess the effect of food on the pharmacokinetics, and safety of Fuzuloparib Capsules in healthy subject.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects over 18 years;
2. Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) of 19.0 to 26.0 kg /m2 (inclusive);
3. Participants should have no fertility plan from signing the informed consent until 6 months after the last dose, and take effective contraceptive measures.

Exclusion Criteria:

1. Subjects with evidence of disease or major surgery;
2. History of drug allergy;
3. Treatment with other investigational drug within 3 months, use of any prescription drugs, Chinese herbal supplements within 4 weeks, and/or need to use any over-the-counter (OTC), food supplements within 2 weeks before the first dose or during the trial;
4. Subjects refuse to stop drinking xanthine-rich beverages or foods at 48 hours before the first dose until the end of the study, and subjects refuse to stop any beverage or food containing grapefruit 7 days before the first dose;
5. Those who have heavy smokers, alcoholics or drug abuse
6. Lactating female subjects or fertile female subjects
7. Those with clinically significant abnormality of physical examination, vital signs and laboratory test during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | day 1 to day 10
Area under the plasma concentration versus time curve from time 0 to last time of measurable concentration (AUC0-t) | day 1 to day 10
Area under the plasma concentration versus time curve from time 0 to infinity (AUC0-∞ ) | day 1 to day 10

SECONDARY OUTCOMES:
The incidence and severity of adverse events/serious adverse events | from ICF signing date to approximate day 23

CONTACTS AND LOCATIONS:
Locations (1):
- Wannan Medical College Yijishan Hospital, Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided